CLINICAL TRIAL: NCT00134550
Title: Improving Diabetic Foot Ulcers With Atorvastatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asker & Baerum Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Odd Erik Johansen, Odd Erik Johansen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The IDUS trial
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Foot Ulcer; Diabetes
Keywords: Diabetes Mellitus; Foot ulcers; Complication; Foot Ulcer, Diabetic
MeSH Terms: conditions — Foot Ulcer; Diabetes Mellitus; Diabetic Foot | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Atorvastatin (10 mg or 80 mg)

SUMMARY:
Lower limb complications are a substantial matter in the diabetic population and studies show that the annual incidence of foot ulcers ranges from 1.0-4.1% while the cumulative lifetime incidence is approximately 15%. Foot ulcers may become complicated by infection or gangrene, and ultimately result in amputation. In addition, foot ulcers have a significant impact on quality of life (QoL). The treatment of diabetic foot ulcers has not made substantial progress in recent years with regards to improved healing although there have been several actions taken to update the process. The current practice consists of wound debridement, treatment of underlying infections and pressure relief. This trial investigates the adjunctive effects of high (80 mg) or low (10 mg) dose atorvastatin to conventional treatment on the healing of diabetic foot ulcers.

DETAILED DESCRIPTION:
The diabetic foot ulcer etiology is multiplex and the wound healing is often not very successful due to various reasons. The ulcer's etiology is associated with peripheral vascular disease, autonomic neuropathy and endothelial. There may also be present some metabolic conditions that are not optimal for wound-healing, delaying the process even more (hyperglycemia, hyperlipidemia, hyperinsulinemia, pro-coagulative state).

It has been shown that statins may improve these aspects making the use of this as adjuvant therapy in treating diabetic foot ulcers an interesting theory. There is so far not any direct evidence for this, although documentation exists for several other possible associated conditions.

This study aims to elucidate the pleiotropic effects of atorvastatin on the healing of diabetic foot ulcers.

Material and Methods:

This 26-week prospective randomised, open, study will be conducted as a pilot to assess the efficacy of atorvastatin in improving diabetic foot-ulcer healing. Atorvastatin will be given in two dosages (10 mg and 80 mg) and evaluations between these groups will be done with regards to improvement in foot ulcer healing, microcirculation and inflammatory markers.

We aim to include 24 patients with diabetes (both type 1 and 2), over the age of 30, of both genders who have a wound duration of less than 12 months. The patients will be recruited from the diabetic out-patient clinics in two centers (Sarpsborg Hospital and Asker and Baerum Hospital).

Study Plan:

We plan to begin the enrolment of eligible patients in autumn 2004. We plan for a 18 month inclusion period and hope to conclude this pilot study by autumn 2006. Results from the study will be presented in international papers or meetings concerning diabetes and complications.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a written informed consent at the enrolment visit
* Men or women above 30 years of age
* Fertile women need to take contraceptives or have to be sterilised
* Diagnosed with any diabetes mellitus type 1 or type 2
* Present foot ulcer with an ulcer duration <= 12 months

Exclusion Criteria:

* Intolerance to statins at any time in the past.
* Unwillingness to participate
* A history of alcohol or drug abuse within the last 2 years
* Foot ulcer with the etiology from vasculitis, pyoderma gangrenosum, angiodermatitis necroticans (hypertensive ulcer), necrobiosis lipoidica, hydrostatic pressure/venous insufficiency or any neoplasms (basalioma, kaposis sarcoma, squamous cell carcinoma etc).
* History of drug-induced hepatitis or previous liver enzyme elevations (> 3 times the upper limit of normal) while taking statins.
* History of drug-induced creatine phosphokinase (CPK) > 3 times the upper limit of normal.
* Critical limb ischemia that requires re-vascularisation procedures within 2 months
* Brachial-ankle index < 0.5
* Other serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the patient's safety or successful participation in the trial.
* Any clinically significant abnormality identified in the enrolment medical history, physical examination, laboratory test which, in the judgement of the investigator, would preclude safe completion of the study.
* Active liver disease or hepatic dysfunction defined as ALAT or ASAT elevations > 2 times the upper limit of normal or total bilirubin > 1.5 times the upper limit of normal.
* Pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of atorvastatin in patients with foot ulcers and type 1 or type 2 diabetes mellitus receiving conventional foot ulcer treatment in improving foot ulcer treatment with regards to completely healed DFU, recurrence of DFU or novel DFU | 26 weeks
Time to complete healing (during 26 weeks of study) | 26 weeks
Recurrence rate of foot ulcers (during 26 weeks of study) | 26 weeks

SECONDARY OUTCOMES:
To assess the efficacy of atorvastatin in patients with foot ulcers and type 1 or type 2 diabetes mellitus receiving conventional foot ulcer treatment in improving: lipid variables and micro-CRP | 26 weeks
Cost of DFU treatment from debut to healing (IDUS substudy) | 2008

CONTACTS AND LOCATIONS:
Overall Officials: Odd E Johansen, MD, Study Chair — Asker and Baerum Hospital
Locations (2):
- Norway (2):
  - Asker and Baerum Hospital, Rud
  - Østfold County Hospital, Sarpsborg

REFERENCES:
- [Result] Johansen OE, Birkeland KI, Jorgensen AP, Orvik E, Sorgard B, Torjussen BR, Ueland T, Aukrust P, Gullestad L. Diabetic foot ulcer burden may be modified by high-dose atorvastatin: A 6-month randomized controlled pilot trial. J Diabetes. 2009 Sep;1(3):182-7. doi: 10.1111/j.1753-0407.2009.00031.x. Epub 2009 Jun 2. PMID 20923537
- See also: EASD — http://www.easd.org/easdwebfiles/annualmeeting/44thmeeting/Posters.pdf